CLINICAL TRIAL: NCT04640519
Title: Telehealth After Stroke Care (TASC): Integrated Multidisciplinary Access to Post-stroke Care
Brief Title: Telehealth After Stroke Care: Integrated Multidisciplinary Access to Post-stroke Care
Acronym: TASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Imama A. Naqvi, Assistant Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAT2612; UL1TR001873 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Health Care Acceptability; Hypertension
Keywords: Telehealth; Blood Pressure (BP)
MeSH Terms: conditions — Stroke; Patient Acceptance of Health Care; Hypertension

STUDY DESIGN:
Intervention Model Description: Multidisciplinary Team Nursing: transitions of care, motivational interview w/ tailored infographics
  Pharmacy: medication education, adherence and titration
  Physician: patient tailored risk factor control, post stroke complications
  Integrated Approach: Home BP monitoring with remote support, Telehealth visits by each discipline, Tailored BP infographics, Patient Reported Outcomes (PROs)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASC Intervention (Experimental): TASC patients will receive a BP monitoring kit and electronic tablet and tailored infographics, and attend 5 telehealth visits over 3 months, including primary care nurse practitioner, pharmacy and stroke neurologist.
  Interventions: Other: TASC intervention
- TASC Control (Active Comparator): Usual care patients will be seen by a primary care nurse practitioner and a stroke neurologist.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Usual care patients will be seen by a primary care nurse practitioner and a stroke neurologist.
  Arms: TASC Control
Other: TASC intervention — TASC patients will receive a BP monitoring kit and electronic tablet with patient tailored BP infographics. They will be scheduled with 5 telehealth visits over 3 months, including primary care nurse practitioner, pharmacy and stroke neurologist.
  Arms: TASC Intervention

SUMMARY:
The Telehealth After Stroke Care (TASC) trial is a pilot randomized controlled trial. It aims to evaluate the feasibility of a telehealth based model providing multidisciplinary access including nursing, pharmacy and physician care, and obtain preliminary evidence of efficacy of an integrated telehealth approach to blood pressure management after stroke.

DETAILED DESCRIPTION:
Hypertension is the most modifiable risk factor for recurrent stroke. Blood pressure (BP) reduction is associated with decreased risk of stroke recurrence but remains poorly controlled in most survivors. Minority groups have a higher prevalence of uncontrolled BP and higher rates of stroke. Limited access contributes to challenges in post-stroke care. Telehealth After Stroke Care (TASC) will be a telehealth intervention that integrates remote BP monitoring and telehealth visits to enhance BP control and promote self-efficacy, with a multidisciplinary approach to improve clinical processes and health outcomes. The investigators will assess for feasibility and obtain preliminary evidence of efficacy. Fifty (50) eligible patients will be screened for inclusion prior to hospital discharge and randomized to TASC or usual care. TASC patients will receive a BP monitoring kit and electronic tablet. They will be scheduled with 5 telehealth visits over 3 months, including primary care nurse practitioner, pharmacy at 4 and 8 weeks and stroke neurologist. Usual care patients will be seen by a primary care nurse practitioner at 1-2 weeks and a stroke neurologist at 1 and 3 months. Data will be collected at 0 and 3 months. The primary outcome will be BP control (BP <140/90 mmHg) at 3 months. The secondary outcome will be self-efficacy in medication adherence and treatment. Interdisciplinary team competency, fidelity, and telehealth satisfaction surveys will be administered. Patient reported outcomes including depression, cognitive function, and socioeconomic determinants will also be collected. Integrated team-based interventions are needed to improve BP control and reduce racial disparities in post-stroke care. It may be feasible and effective in enhancing post-stroke BP control and promoting self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of hypertension (by clinical history or hospital BP ≥140/90 on two occasions)
* Plan for discharge home after stroke
* Ability to provide consent (patient or caregiver)

Exclusion Criteria:

* Modified Rankin scale ≥ 4 at time of enrollment (severely disabled)
* Pregnancy
* Severe psychiatric illness
* Dialysis or diagnosis of end stage renal disease
* Life expectancy < 1 year or terminal illness
* Symptomatic flow limiting cerebrovascular stenosis without plan for intervention, or long-term BP goal ≥ 140/90

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imama Naqvi, MD, Principal Investigator — Columbia University
Locations (1):
- The Neurological Institute of New York, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naqvi IA, Cheung YK, Strobino K, Li H, Tom SE, Husaini Z, Williams OA, Marshall RS, Arcia A, Kronish IM, Elkind MSV. TASC (Telehealth After Stroke Care): a study protocol for a randomized controlled feasibility trial of telehealth-enabled multidisciplinary stroke care in an underserved urban setting. Pilot Feasibility Stud. 2022 Apr 11;8(1):81. doi: 10.1186/s40814-022-01025-z. PMID 35410312
- [Derived] Naqvi IA, Strobino K, Kuen Cheung Y, Li H, Schmitt K, Ferrara S, Tom SE, Arcia A, Williams OA, Kronish IM, Elkind MSV. Telehealth After Stroke Care Pilot Randomized Trial of Home Blood Pressure Telemonitoring in an Underserved Setting. Stroke. 2022 Dec;53(12):3538-3547. doi: 10.1161/STROKEAHA.122.041020. Epub 2022 Oct 31. PMID 36314123

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TASC Intervention | TASC Control
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TASC Intervention | TASC Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (15.6) | 62.6 (12.4) | 64.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 5 | 5 | 10
  Non-Hispanic Black | 6 | 10 | 16
  Dominican / Hispanic | 14 | 8 | 22
  Non-Hispanic Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 139.7 (18.9) | 142.0 (18.9) | 140.9 (18.8)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 80.2 (10.5) | 79.9 (11.8) | 80.1 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Systolic BP Control
Description: The outcome of BP control will be defined by change in mean awake systolic blood pressure from baseline at the time of discharge through remote monitoring at 3 months to be < 130 mmHg. BP control will be determined by the mean 24-hr blood pressure through remote monitoring at 3 months and survey patient reported outcomes for all participants.
Time Frame: Up to 3 months
Population: Only data of evaluable participants were included in the analysis: 21 out of 25 TASC Intervention patients and 16 out of 25 TASC Control patients.
Measure: Number; unit: percentage of participants
Arm/Group | TASC Intervention | TASC Control
Number analyzed (Participants) | 21 | 16
percentage of participants | 76 | 25

2. Primary Outcome: Percentage of Participants Who Completed at Least 1 Video Visit
Description: This measures the feasibility of the TASC model, the interdisciplinary team competency, fidelity of implementation.
Time Frame: 3 months
Population: Only data of evaluable participants were included in the analysis: 23 out of 25 TASC Intervention patients and 24 out of 25 TASC Control patients.
Measure: Number; unit: percentage of participants
Arm/Group | TASC Intervention | TASC Control
Number analyzed (Participants) | 23 | 24
percentage of participants | 91 | 75

3. Secondary Outcome: Medication Adherence Percentage
Description: Feasibility as assessed by patient reported outcomes of self-efficacy in bp medication adherence after study intervention.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TASC Intervention | TASC Control
Number analyzed (Participants) | 21 | 16
percentage of participants | 67 | 63

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | TASC Intervention | TASC Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT04640519/Prot_SAP_000.pdf